CLINICAL TRIAL: NCT03413787
Title: The Türkish Version of the Freezing of Gait Questionnaire in Patients With Parkinson's Disease
Brief Title: The Türkish Version of the Freezing of Gait Questionnaire
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Sevim ACARÖZ CANDAN, Head of the Department of Physiotherapy and Rehabilitation, Ordu University
Other Study IDs: Ordu2
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Parkinson Disease; Motor Disorder; Gait Disorders, Neurologic
MeSH Terms: conditions — Parkinson Disease; Motor Disorders; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The freezing of gait (FOG) is one of the disabling symptoms in Parkinson's disease. The diagnosis and assessment of the FOG may be diffucult, but it is absolutely necessary. The aim of this study was to develop a Türkish version of the freezing of gait questionnaire (FOG-Q) and assess the validity and reliability of this Türkish version.

The researchers firstly communicated with the developers of the FOG-Q. The permission for Turkish version was received by Giladi. Then, the FOG-Q will be adapted into Türkish using forward-backward translation by three native Türkish-speaking forward translators and one native English-speaking backward translator. The internal reliability of the FOG-Q Türkish version will be assessed using Cronbach's alpha, and item analyses will be conducted by examining the effect on Cronbach's alpha of excluding each of the six FOG-Q items individually. The test-retest reliability will be assessed using intraclass correlation coefficient (ICC).

Convergent validity will be evaluated by means of Spearman rank correlation coefficient (rs). In this section will be determined the correlation between the FOG-Q scores and scores of the UPDRS motor section , Berg Balance Scale, Timed up and go test, Falls Efficacy Scale and Hoehn and Yahr stages.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of idiopathic PD
* able to walk with or without a walking device

Exclusion Criteria:

* a diagnosis of other neurological disorders
* any other medical conditions
* not able to take commands.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be selected from neurologic clinic.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Türkish version of the Freezing of Gait Questionnaire | 5 minutes
  Türkish version of the Freezing of Gait Questionnaire determine the episode of the freezing and the severity of the freezing by six items. Each items with five response categories (scored from 0 to 4) that are summed into a total score (range 0-24; higher scores = more severe FOG).

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale-part III | 5 minutes
  Türkish version of the Unified Parkinson's Disease Rating Scale (UPDRS) will be used. UPDRS-part III evaluate the motor symptoms observational by neurologist. (UPDRS) scored from 0 (normal) to 4 (maximum disability); the total score change between 0 and 56. High scores mean worse motor function.
Berg Balance Scale | 10 minutes
  The balance will be evaluated observational during 14 different balance activities. Each item will be scored between 1 and 4. The test score change between 0 and 56. The high score indicates better balance ability.
Timed up and go test | 2 minutes
  This test will be used to measure the progress of balance, sit to stand, and walking. The participants stands up upon therapist's command walks 3 meters, turns around, walks back to the chair and sits down.
  The time stops when the patient is seated. Time will be recorded.
Fall Efficacy Scale | 5 minutes
  7 item-Fall Efficacy Scale (FES) will be used. FES is a questionnaire that assesses fear of falling. The score of the scale change 0-100 and the score above 70 indicates the fear of falling.
Hoehn and Yahr Scale | 2 minutes
  The Hoehn and Yahr Scale (HYS) will be used to assess the severity in Parkinson's Disease based on clinical findings and functional disability. In HYS is a rating scale measured in an ordinal level. Here higher rates describe an increase severity of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim ACARÖZ CANDAN, PhD, Principal Investigator — Ordu University
Locations (1):
- Sevim ACARÖZ CANDAN, Ordu, Altinordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No